CLINICAL TRIAL: NCT04106063
Title: A New Speech, Spatial, and Qualities of Hearing Scale Short-Form for Deaf Children
Acronym: KID SSQ12
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0533
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Deafness; Pediatric
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- deaf children: All Children between 7 and 17 years old attending medical appointment for temporary or persistent deafness in our Ear, Nose and Throat (ENT) department
  Interventions: Other: KID SSQ12 questionnaire

INTERVENTIONS:
Other: KID SSQ12 questionnaire — During a face to face interview (maximum 15 minutes), the child will complete a short questionnaire (KID SSQ12 questionnaire) to assess his auditory difficulties

SUMMARY:
Deafness significantly affects several auditory tasks of everyday life in children: understanding speech in quiet and noisy environments, spatial location of sounds ...

These difficulties in locating sound sources are often ignored by parents and underestimated by children. Nowadays we there is specific tools to evaluate these problems in children. Indeed, there is a validated French questionnaire (Speech and Spatial Questionnaire SSQ) for adults that evaluates auditory abilities, including sound localization, in different tasks of daily life. Although robust, this questionnaire includes 49 questions and is too long for daily use in consultation. For this reason, Moulin et al validated in 2018 a short version of the SSQ questionnaire for adults with only 15 items.

Based on this model, the aim of this study is to develop and test a paediatric questionnaire with 12 items to assess more specifically auditory difficulties in deaf children. This questionnaire will follow the validated frame of the adult SSQ questionnaire and will consist of three subscales: speech hearing (4 items), spatial hearing (4 items), and qualities of hearing (4 items). These 3 subscales are identical to those defined in long and short form pf the adult SSQ questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 7-17 (inclusive)
* Attending medical appointment for temporary or persistent deafness
* Able to understand the experimental instructions

Exclusion Criteria:

none-

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All Children between 7 and 17 years old attending medical appointment for temporary or persistent deafness in our ENT department
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
KID SSQ12 questionnaire score | At inclusion
  This questionnaire evaluates auditive abilities (including sound localisation) in different every day life tasks, in deaf children. It is made up of 12 items ; for each item the score range is between 0 (worse outcome) and 10 (best outcome). The questionnaire is devided into 3 subscores of 4 items : speech audition, spatial audition and quality of audition.
  Thanks to that tool, internal structures (internal consistency, sub-scale structure obtained by principal component analysis and cluster analysis) and psychometric values will be compared with adult versions of the questionnaire (complete and abbreviated) published in the international literature. Overall scores, scores by subscales and items will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Eric TRUY, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- ENT departement, Edouard Herriot Hospital, Lyon, France